CLINICAL TRIAL: NCT06667622
Title: Sodium Glycididazole Reduces Chemoradiotherapy-related Adverse Reactions During Concurrent Chemoradiotherapy for Locally Advanced Non-small Cell Lung Cancer
Brief Title: Sodium Glycididazole Reduces the Adverse Reactions of Concurrent Chemoradiotherapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC4420
Record Dates: First submitted 2024-09-22; First posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-08

CONDITIONS: Chemoradiotherapy
MeSH Terms: interventions — sodium glycididazole; Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (1):
- Sodium glycididazole combined with concurrent chemoradiotherapy group (Experimental): Patients with unresectable locally advanced non-small cell lung cancer after neoadjuvant chemoradiotherapy are treated with sodium glycididazole during concurrent chemoradiotherapy.
  Interventions: Drug: sodium glycididazole

INTERVENTIONS:
Drug: sodium glycididazole — Sodium glycididazole is intravenously infused at a dose of 800mg at 60 min before radiotherapy and used on Mondays, Wednesdays and Fridays during radiotherapy.
  Other Names: Sodium glycididazole combined with concurrent chemoradiotherapy

SUMMARY:
To evaluate the efficacy and toxicity of sodium glycididazole combined with concurrent chemoradiotherapy in patients with unresectable locally advanced non-small cell lung cancer after neoadjuvant chemoradiotherapy.

DETAILED DESCRIPTION:
1. To evaluate the efficacy and toxicity of concurrent chemoradiotherapy combined with sodium glycididazole in patients with unresectable locally advanced non-small cell lung cancer after neoadjuvant chemoradiotherapy, and to explore sodium glycididazole as a new way to inhibit the occurrence of radiation esophagitis and reduce the occurrence of radiation pneumonitis and lymphopenia.
2. To evaluate the sensitization effect of sodium glycididazole in the anti-tumor activity during concurrent chemoradiotherapy, as well as the changes in the anti-tumor immune response in peripheral blood, in order to screen out the dominant population and the predictive biomarkers with fewer related toxic and side effects.
3. By exploring the correlation between the expression level of NLRP3 inflammasome activation related molecules and imaging changes in peripheral blood after radiotherapy and the toxicity of radiotherapy and chemotherapy, a risk model for predicting radiation esophagitis after concurrent radiotherapy and chemotherapy for non-small cell lung cancer was further constructed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed non-small cell lung cancer.
2. Patients with unresectable stage II-III non-small cell lung cancer after neoadjuvant therapy.
3. ECOG PS 0-2
4. Adequate organ and bone marrow function.

Exclusion Criteria:

1. History of previous radiotherapy.
2. The previous immune-related pneumonitis ≥ grade 2.
3. Local lesions require surgery.
4. History of another primary malignancy.
5. History of active primary immunodeficiency.
6. Histological findings showed mixed small cell lung cancer and non-small cell lung cancer.
7. For any unmitigated toxicity during pre-study chemoradiotherapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-29 (Actual); Primary Completion 2026-01-10 (Estimated); Study Completion 2026-07-20 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of grade 3 and above radiation esophagitis | 8 weeks
  Radiation esophagitis of grade 3 or higher is graded according to the toxicity criteria of the CTCAE v5.0.
Incidence and severity of grade 2 and above radiation pneumonitis | 8 weeks
  Radiation pneumonitis of grade 2 or higher is graded according to the toxicity criteria of the CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Deng, MD, Study Chair — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No